CLINICAL TRIAL: NCT04860544
Title: Red Blood Cell Transfusion and Its Association With Vascular Pedicle Thrombosis
Brief Title: Is Red Blood Cell Transfusion a Risk Factor for Vascular Pedicle Thrombosis? The Study Case of a Latin American Cohort
Acronym: RBCT
Status: Completed | Type: Observational
Sponsor: Fundación Universitaria de Ciencias de la Salud (Other)
Collaborators: Hospital de San Jose (Other)
Responsible Party: Sponsor
Other Study IDs: 462-3762-17
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Vascular Thrombosis
Keywords: Free flap; Thrombosis; Blood transfusion
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: RED BLOOD CELLS TRANFUSION

SUMMARY:
The present cohort was performed between January of 2014 and December of 2019. It included 302 free flaps conducted between January 2006 and December 2019 in the Hospital de San José and Hospital Infantil Universitario de San José in Bogotá, Colombia. Its aims were to determine whether there is an association between perioperative red blood cell transfusion and the risk of free flap vascular pedicle thrombosis. The exposure was the red blood cell transfusion therapy during the perioperative eriod, and the primary outcome was the occurrence of vascular pedicle thrombosis, which was defined as the intraoperative visualization of arterial or venous thrombosis of the vascular pedicle observed until seven days following the procedure.

As a secondary outcome, the presence of clinical signs of arterial or venous flap suffering. Red blood cell transfusion was prescribed by the attending anesthesiologist.

The methodology included data collection from medical records history, statistical analysis (incidence of thrombosis and to plot survival curves, the incidence rates calculated for every 1000 free flaps and the analysis between thrombosis and perioperative variables) by Kaplan Meier method and Cox regression models and its interpretation. The results showed that red blood cell transfusion during the perioperative period did not represent a risk for vascular pedicle thrombosis and also discarded a possible effect on the free flap survival.

DETAILED DESCRIPTION:
The study included patients who underwent free flap surgery between January 2006 and December 2019 in the Hospital de San José and Hospital Infantil Universitario de San José in Bogotá, Colombia. Criteria for exclusion were history of deep vein thrombosis, pulmonary embolism, systemic lupus erythematosus, antiphospholipid syndrome, hypercoagulability syndrome, and previous medication with oral or parenteral anticoagulant within the past year of the surgery. A standardized Google App for Work form was created where participant's medical records were registered. The exposure criteria were RBCT, and the primary outcome was the occurrence of VPT, which was defined as the intraoperative visualization of arterial or venous thrombosis in the vascular pedicle, observed up until seven days after the procedure. As a secondary outcome, the presence of clinical signs of arterial flap suffering (pallor, decreased capillary filling time, decreased skin turgor, , venous congestion: blue dermal bleeding, and poikilothermia). As well as the absence of blood flow measured by Doppler ultrasound that was registered from the beginning until the outcome. Different clinical characteristics were recorded such as: age, gender, body mass index (BMI), diabetes (fasting blood glucose >126 mg/dl or random glucose value >200 mg/dl), arterial hypertension (persistently high value >140/90 mmHg or use of antihypertensive medication for adequate control) anesthetic risk (ASA Classification), most recent pre-surgical hemoglobin (Hb mg/dl), most recent pre-surgical hematocrit (Ht %), anemia (Hb <12mg/dl or Hto <36% in children under 14 and women of childbearing age, Hb <13 mg/dl or Hto <39% in men over 14 or postmenopausal women), history of chemotherapy during the past year, history of radiation therapy in the flap donor or free flap recipient site In regard to the surgery performed, the following variables were analyzed: indication of procedure, free flap donor site, free flap recipient site, type of flap, whether or not other concomitant surgical procedures were being performed (oncological resections, osteosynthesis, tumor resections) and intra-operative bleeding according to the records from anesthesiologists' evaluations. The information was exported from the standardized formats to a database for statistical analysis through statistical packages R and Stata 15® licensed by the Fundación Universitaria de Ciencias de la Salud - FUCS.

The exposed group corresponded to patients who received red blood cell transfusion during the perioperative period of free flap surgery (defined as: 24 hours before, during and up to 24 hours after the procedure).

- The unexposed group corresponded to patients who did not receive red blood cell transfusion during the perioperative period of free flap surgery (defined as: 24 hours before, during and up to 24 hours after the procedure).

ELIGIBILITY:
Inclusion Criteria:

* The study included patients who underwent free flap surgery between January 2006 and December 2019 in the Hospital de San José and Hospital Infantil Universitario de San José in Bogotá, Colombia.

Exclusion Criteria:

* Criteria for exclusion were history of deep vein thrombosis, pulmonary embolism, systemic lupus erythematosus, antiphospholipid syndrome, hypercoagulability syndrome and previous medication with oral or parenteral anticoagulant within the past year of the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent free flap surgery between January 2006 and December 2019 in the Hospital de San José and Hospital Infantil Universitario de San José in Bogotá, Colombia
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
VASCULAR PEDICLE THROMBOSIS | 7 DAYS
  the primary outcome was the occurrence of VPT, which was defined as the intraoperative visualization of arterial or venous thrombosis of the vascular pedicle observed until seven days following the procedure

SECONDARY OUTCOMES:
arterial or venous non-thrombotic vascular complications in the flap | 7 DAYS
  As a secondary outcome, the presence of clinical signs of arterial flap suffering (pallor, decreased capillary filling time, decreased skin turgor, scarce dermal bleeding and poikilothermia) or venous flap suffering (cutaneous cyanosis, increased turgor, venous congestion: blue dermal bleeding, and poikilothermia). As well as the absence of blood flow measured by Doppler ultrasound was registered from the beginning until the outcome

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS E TORRES FUENTES, MD.PS, Principal Investigator — FUNDACION UNIVERSITARIA DE CIENCIAS DE LA SALUD

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill JB, Patel A, Del Corral GA, Sexton KW, Ehrenfeld JM, Guillamondegui OD, Shack RB. Preoperative anemia predicts thrombosis and free flap failure in microvascular reconstruction. Ann Plast Surg. 2012 Oct;69(4):364-7. doi: 10.1097/SAP.0b013e31823ed606. PMID 22964664
- [Result] Kroll SS, Schusterman MA, Reece GP, Miller MJ, Evans GR, Robb GL, Baldwin BJ. Choice of flap and incidence of free flap success. Plast Reconstr Surg. 1996 Sep;98(3):459-63. doi: 10.1097/00006534-199609000-00015. PMID 8700982
- [Result] Nakatsuka T, Harii K, Asato H, Takushima A, Ebihara S, Kimata Y, Yamada A, Ueda K, Ichioka S. Analytic review of 2372 free flap transfers for head and neck reconstruction following cancer resection. J Reconstr Microsurg. 2003 Aug;19(6):363-8; discussion 369. doi: 10.1055/s-2003-42630. PMID 14515225
- [Result] Novakovic D, Patel RS, Goldstein DP, Gullane PJ. Salvage of failed free flaps used in head and neck reconstruction. Head Neck Oncol. 2009 Aug 21;1:33. doi: 10.1186/1758-3284-1-33. PMID 19698095
- [Result] Zhou W, Zhang WB, Yu Y, Wang Y, Mao C, Guo CB, Yu GY, Peng X. Risk factors for free flap failure: a retrospective analysis of 881 free flaps for head and neck defect reconstruction. Int J Oral Maxillofac Surg. 2017 Aug;46(8):941-945. doi: 10.1016/j.ijom.2017.03.023. Epub 2017 Apr 14. PMID 28416356
- [Result] Cannady SB, Hatten KM, Bur AM, Brant J, Fischer JP, Newman JG, Chalian AA. Use of free tissue transfer in head and neck cancer surgery and risk of overall and serious complication(s): An American College of Surgeons-National Surgical Quality Improvement Project analysis of free tissue transfer to the head and neck. Head Neck. 2017 Apr;39(4):702-707. doi: 10.1002/hed.24669. Epub 2016 Dec 21. PMID 28000297
- [Result] Heidekrueger PI, Ninkovic M, Heine-Geldern A, Herter F, Broer PN. End-to-end versus end-to-side anastomoses in free flap reconstruction: single centre experiences. J Plast Surg Hand Surg. 2017 Oct;51(5):362-365. doi: 10.1080/2000656X.2017.1283321. Epub 2017 Feb 2. PMID 28151027